CLINICAL TRIAL: NCT03154879
Title: Prospective Multi-center Study to Verify Neurological Prognostic Value of Amplitude-integrated Electroencephalogram in Cardiac Arrest Patients Treated With Therapeutic Hypothermia
Brief Title: Frontal Amplitude-integrated Electroencephalogram in Early Prognostication After Cardiac Arrest
Acronym: FRONTEER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Kyu Nam Park, Professor, Seoul St. Mary's Hospital
Other Study IDs: 2017-CMC-07
Record Dates: First submitted 2017-05-07; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Heart Arrest
Keywords: Heart arrest; Hypothermia; EEG; Prognosis
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Comatose cardiac arrest survivors
  Interventions: Device: Amplitude integrated electroencephalography

INTERVENTIONS:
Device: Amplitude integrated electroencephalography — Frontal Amplitude-integrated Electroencephalogram in Early Prognostication After Cardiac Arrest

SUMMARY:
The investigators examine the prognostic value of continuous electroencephalography on frontal area of brain according to time by performing amplitude-integrated electroencephalography (aEEG) on cardiac arrest patients receiving therapeutic hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* age: 19 years and older
* underwent TH

Exclusion Criteria:

* Died within 72 h after cardiac arrest
* Spontaneous or traumatic brain injury
* Known history of neurological diseases (such as epilepsy)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose cardiac arrest survivors treated with TH
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of time to normal trace to good neurological outcome evaluated by cerebral performance category (CPC) score 1 to 2 | at day 180
  Time to normal trace is defined as time to regained normal trace on aEEG after return of spontaneous circulation.
  The normal trace is defined as continuous cortical activity on the raw EEG scan; in addition, the upper margin of the aEEG scan, referred to as the aEEG maximum, was >10 uV, and the lower margin of the aEEG scan, referred to as the aEEG minimum, was >5 uV.

SECONDARY OUTCOMES:
Comparison of time to normal trace to poor neurological outcome evaluated by CPC score 3 to 5 | at day 180
  Time to normal trace is defined as time to regained normal trace on aEEG after return of spontaneous circulation.
  The normal trace is defined as continuous cortical activity on the raw EEG scan; in addition, the upper margin of the aEEG scan, referred to as the aEEG maximum, was >10 uV, and the lower margin of the aEEG scan, referred to as the aEEG minimum, was >5 uV.
Comparison of unfavorable aEEG patterns to poor neurological outcome evaluated by CPC score 3 to 5 | at day 180
  Unfavorable aEEG patterns include flat trace (FT), burst-suppression (BS) and status epilepticus (SE).
  FT is defined as isoelectric activity. BS is defined as the virtual absence of activity (<2uV) between bursts of high voltage (>25 uV).
  SE was defined as repetitive epileptiform discharges with amplitudes >50 uV and a median frequency 1 Hz for >30 min.
Comparison of diffusion weighted image (DWI) to poor neurological outcome evaluated by CPC score 3 to 5 | at day 180
Comparison of the levels of serum neuron specific enolase (NSE) to poor neurological outcome evaluated by CPC score 3 to 5 | at day 180
Comparison of convulsive movement and electrical status epilepticus (SE) to poor neurological outcome evaluated by CPC score 3 to 5 | at day 180

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Nam Park, MD, Study Chair — Seoul St. Mary's Hospital
Locations (4):
- South Korea (4):
  - Samsung Changwon Hospital, Changwon
  - Chonnam National University, Gwangju
  - Seoul St. Mary's hospital, Seoul
  - KEPCO Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Web based Case Report Form